CLINICAL TRIAL: NCT03094247
Title: Improved Polyunsaturated Ready-to-use Therapeutic Food for Improved Neurocognitive Outcomes in Severe Acute Malnutrition
Brief Title: Feeding Malnourished Children Different Types of Fatty Acids to Promote Neurocognitive Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Texas at Austin (Other); Cornell University (Other); Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMPUFA17
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Severe Acute Malnutrition
Keywords: Malnutrition; Micronutrients; Polyunsaturated fatty acids; Ready-to-use therapeutic foods; Omega-3 fatty acids; Peanuts
MeSH Terms: conditions — Severe Acute Malnutrition; Malnutrition | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional RUTF (S-RUTF) (Active Comparator): This is the control group for the study, which will receive the international standard of care therapeutic food. S-RUTF is made with conventional peanuts, which are inherently high in omega-6 linoleic acid.
  Interventions: Drug: Amoxicillin; Dietary Supplement: S-RUTF
- High oleic RUTF (HO-RUTF) (Experimental): The treatment provided to children randomized to this arm of the study includes nutritional content comparable to S-RUTF with the exception of a low lineoleic acid/high oleic acid ratio formulated with high oleic content peanuts.
  Interventions: Drug: Amoxicillin; Dietary Supplement: HO-RUTF
- DHA-supplemented HO-RUTF (D-HO-RUTF) (Experimental): The treatment provided to children randomized to this arm of the study mirrors that provided by HO-RUTF with that addition of supplemental DHA at a level higher than attainable with optimal precursors.
  Interventions: Drug: Amoxicillin; Dietary Supplement: D-HO-RUTF

INTERVENTIONS:
Drug: Amoxicillin — All patients with severe acute malnutrition will receive a course of amoxicillin.
  Other Names: Amoxil
Dietary Supplement: HO-RUTF — HO-RUTF: Milk, perilla oil, palm oil, white sugar, high oleic peanuts
  Arms: High oleic RUTF (HO-RUTF)
Dietary Supplement: D-HO-RUTF — D-HO-RUTF: DHA, milk, perilla oil, palm oil, white sugar, high oleic peanuts
  Arms: DHA-supplemented HO-RUTF (D-HO-RUTF)
Dietary Supplement: S-RUTF — S-RUTF: Milk, canola oil, palm oil, white sugar, standard peanuts
  Arms: Conventional RUTF (S-RUTF)

SUMMARY:
An appropriate balance of omega-6 and omega-3 fatty acids is important for support of neurocognitive development in healthy infants and toddlers. In young children recovering from severe acute malnutrition (SAM), excess omega-6 intake depletes omega-3 fatty acid status. This research will evaluate how novel ready-to-use therapeutic foods (RUTF) with balanced fatty acids improve the metabolic and neurocognitive effects in young children in Malawi recovering from SAM, yielding new knowledge that also has implications for development of well-nourished children.

ELIGIBILITY:
Inclusion Criteria:

* 6-59 months
* An acceptable appetite defined by the ability to consume 30 grams RUTF within 20 minutes
* Mid Upper Arm Circumference <11.5 cm, weight-for-height z-score < -3, or bilateral pitting edema on the dorsum of the feet

Exclusion Criteria:

* Participation in any other ongoing study or supplementary feeding program
* Children with a chronic medical condition, including cerebral palsy, static encephalopathy, congenital heart disease, gastrointestinal disease, or peanut allergy

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2897 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Neurocognitive outcome | Time Frame: 4 to 7 months after nutritional outcome
  Measured by score on the Malawian Developmental Assessment Test (MDAT). The scale is continuous and interval in nature, the range varies by population
  * The scale title is "Malawi Developmental Assessment Tool z-score"
  * The primary outcome is Global z-score, titled "Global z-sore"
  * Secondary outcomes are 4 sub-domain z-scores are titled "Gross motor z-score", "Fine motor z-score", Language z-score", and "Social z-score"
Neurocognitive outcome | Time Frame: within 4 weeks after nutritional outcome
  Defined by Willatts intention score adapted for field training, 3 problems to be tested. The scale is ordinal in nature, with higher values indicated better scores
  * The scale title is "Intention Score"
  * Problem 1 is scored 0 - 4
  * Problem 2 is scored 0 - 4
  * Problem 3 is scored 0 - 8

SECONDARY OUTCOMES:
Nutritional recovery | Up to 12 weeks following enrollment
  Defined by resolution of edema AND mid-upper arm circumference [MUAC] >12.4cm, AND/OR a weight/height z-score [WHZ] >-3
Attentional orienting speed | 4-7 months after nutritional after nutritional outcome
  Measured by mean saccade latency to peripheral targets
Adverse Events | Fortnightly follow up visits up to 12 weeks following enrollment
  Measured by number of days diarrhea and/or rashes.
Acceptance of RUTF | Fortnightly follow up visits up to 12 weeks following enrollment
  Mother's report of if the child ate the food well. This is a yes or no question.

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Study Chair — Washington University School of Medicine
Locations (1):
- University of Malawi College of Medicine, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article after deidentification will be indefinitely available within 9 months following article publication through The Washington University Open Scholarship Institutional Repository.
Supporting Information: Study Protocol
Time Frame: Data will be available within 9 months of article publication. Data will remain available indefinitely.
Access Criteria: Anyone who wishes to access the data.
URL: https://openscholarship.wustl.edu/data/101/

REFERENCES:
- [Derived] Stephenson K, Callaghan-Gillespie M, Maleta K, Nkhoma M, George M, Park HG, Lee R, Humphries-Cuff I, Lacombe RJS, Wegner DR, Canfield RL, Brenna JT, Manary MJ. Low linoleic acid foods with added DHA given to Malawian children with severe acute malnutrition improve cognition: a randomized, triple-blinded, controlled clinical trial. Am J Clin Nutr. 2022 May 1;115(5):1322-1333. doi: 10.1093/ajcn/nqab363. PMID 34726694
- Available data/document: Individual Participant Data Set — https://openscholarship.wustl.edu/data/101/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT03094247/Prot_SAP_ICF_000.pdf